CLINICAL TRIAL: NCT04613024
Title: Beneficial Side Effects of Topiramate in Obese Patients Undergoing Total Joint Arthroplasty, a Study of Opiate Consumption and Weight Reduction
Brief Title: Beneficial Side Effects of Topiramate in Obese Patients Undergoing Total Joint Arthroplasty
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Not funded
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Derek Amanatullah, Assistnat professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 56915
Record Dates: First submitted 2020-10-01; First posted 2020-11-03 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Weight Loss; Pain, Postoperative
MeSH Terms: conditions — Weight Loss; Pain, Postoperative | interventions — Topiramate; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experiment (Experimental): Topamax randomized group
  Interventions: Drug: Topamax
- Control (Active Comparator): Gabapentin randomized group
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Topamax — Experiment randomized group will be prescribed Topamax before and after surgery with follow up at regular interval
  Arms: Experiment
Drug: Gabapentin — Control group will be prescribed gabapentin after surgery with follow up at regular interval
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of topiramate (TPM) in obese patients with respect to weight loss and pain after total joint replacement surgery

DETAILED DESCRIPTION:
Investigator hypothesize that low dose peri-operative topiramate is superior to gabapentin in reducing postoperative pain and opioid consumption after primary TJA with a more favorable side effect profile that will facilitate patient optimization via pre- and postoperative weight loss.

ELIGIBILITY:
Inclusion Criteria

* Patient will be eligible for the study if they are scheduled for a primary TKA or THA with a BMI >30 and <40 kg/m2, or >40 kg/m2
* Patients refusing bariatric surgery or having had prior bariatric surgery

Exclusion Criteria

* Patients will be ineligible to participate if they have any of the following:
* known topiramate or gabapentin allergy
* history of seizure disorder
* chronic opiate use pre-operatively
* history of nephrolithiasis
* history of acute angle closure glaucoma
* recurrent major depression
* presence or history of suicidal behavior or ideation with intent to act
* current substantial depressive symptoms (Patient Health Questionnaire total score >10), pregnancy
* child-bearing potential and not on contraception
* age <18 years
* major neurocognitive disorder
* metabolic acidosis
* incarcerated status
* bilateral surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Determine the reduction in Opioid Consumption | 3 months
  Postoperative morphine equivalent opiate use and opiate refill requests after discharge will be compared post randomization to receive one of the two medications for multimodal pain control.
Evaluate the Side Effect Profiles of Topiramate | 3 months
  Perioperative weight change experienced by patients will be compared after randomization to receive one of the two medications. Weight change is measured in lbs
Evaluate the Side Effect Profiles of gabapentin | 3 months
  Perioperative weight change experienced by patients will be compared after randomization to receive one of the two medications. Weight change is measured in lbs

SECONDARY OUTCOMES:
Harris hip score - Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin | 1 week
  Harris hip score will be calculated after randomization at the pre-operative visit. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Harris hip score - Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin at 2 weeks | 2 week
  Harris hip score will be calculated after surgery. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Harris hip score - Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin at 6 weeks | 6week
  Harris hip score will be calculated after surgery. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Harris hip score -Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin at 3 months | 3 months
  Harris hip score will be calculated after surgery. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
SF12- Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin at 3 months | 3 months
  SF12 will be calculated after surgery
SF12 Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin at 2weeks | 2 week
  SF12 will be calculated after surgery
SF12- Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin at 6 weeks | 6 week
  SF12 will be calculated after surgery
SF12- Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin at 1 week | 1 week
  SF12 will be calculated after surgery
WOMAC score Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin at 6 weeks | 6 week
  WOMAC score will be calculated after surgery. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores
WOMAC score - Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin at 2 weeks | 2 week
  WOMAC score will be calculated after surgery. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores
WOMAC score - Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin at 3 months | 3 months
  WOMAC score will be calculated after surgery. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores
WOMAC score - Evaluate Short-term Arthroplasty-related Outcomes and Complications while on Topiramate or Gabapentin at 3 months | 1 week
  WOMAC score will be calculated after surgery. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, United States Minor Outlying Islands